CLINICAL TRIAL: NCT04061577
Title: Transcranial Electrical Stimulation in Stroke EaRly After Onset Clinical Trial_ Bridging and Adjunctive Neuroprotection
Brief Title: Transcranial Direct Current Stimulation as a Neuroprotection in Acute Stroke Before and After Thrombectomy
Acronym: TESSERACT-BA
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Interim Analysis
Sponsor: University of California, Los Angeles (Other)
Collaborators: The City College of New York (Other)
Responsible Party: Principal Investigator, Mersedeh Bahr Hosseini, MD, Principal Investigator, University of California, Los Angeles
Allocation: Randomized | Model: Sequential | Masking: Single | Purpose: Treatment
Other Study IDs: 19-000529
Record Dates: First submitted 2019-07-30; First posted 2019-08-20 (Actual); Results first posted 2023-07-20 (Actual); Last update posted 2023-07-20 (Actual); Status verified 2023-06

CONDITIONS: Acute Ischemic Stroke
Keywords: Transcranial direct current stimulation; Bridging neuroprotection; Adjunctive neuroprotection
MeSH Terms: conditions — Ischemic Stroke | interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Intervention Model Description: Traditional 3+3 (rule-based, modified Fibonacci) dose-escalation design
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (2):
- Stimulation arm (Experimental): Patients will be randomized to active treatment (C-tDCS) vs sham stimulation in a 3:1 ratio. There will be 6 dose tiers:
  Tier 1 - 1 mA, and Tier 2- 2 mA: Consist of a single stimulation cycle (20min) after the endovascular procedure (EVT) in patients with TICI<2c,3 and negative immediate post-EVT CT scan for definitive evidence of ICH.
  Tier 3 - 1 mA and Tier 4- 2mA consist of 2 treatment cycles after the EVT in patients with TICI<2c and 3, and negative immediate post-EVT CT scan for definitive evidence of ICH.
  Tier 5 - 1 mA and tier 6- 2 mA consist of 3 treatment cycles. The first cycle will be up to 20 min cycle, after initial imaging and prior to arterial puncture, the second and third cycles after EVT in patients with TICI<2c and 3 and negative immediate post-EVT CT scan for definitive evidence of ICH.
  Interventions: Device: Transcranial Direct Current Stimulation (tDCS)
- Sham arm (Sham Comparator): Patients in the sham stimulation arm at all the tiers will have the cap and electrodes in place, and sham switch moved but without delivery of electrical stimulation.
  Interventions: Device: Transcranial Direct Current Stimulation (tDCS)

INTERVENTIONS:
Device: Transcranial Direct Current Stimulation (tDCS) — 20 minutes of Cathodal tDCS after +/- before endovascular thrombectomy (EVT)

SUMMARY:
This proposal is a prospective, single-center, dose-escalation safety, tolerability, feasibility and potential efficacy study of transcranial direct current stimulation (tDCS) in acute stroke patients with substantial salvageable penumbra due to a large vessel occlusion before and after endovascular therapy.

DETAILED DESCRIPTION:
This is a single-center, sham-controlled, dose-escalation study where cathodal tDCS is delivered to threatened but not yet irreversibly damaged (penumbral) tissue in patients with large vessel occlusion who are undergoing recanalization procedure. Patients will be randomized in a 3:1 design, to cathodal versus sham (control) stimulation, at each six designed dose tiers. The dose tiers will be increasing in both intensity and duration of the stimulation. All patients will be receiving the first dose (stimulation cycle) after the recanalization procedure and patients at dose tiers 5-6 will also be receiving stimulation cycles before the recanalization procedure begins.

The occurrence of symptomatic intracranial hemorrhage will determine the pace of the escalation through the dose tiers.

ELIGIBILITY:
Inclusion criteria

* New focal neurologic deficit consistent with AIS
* Age≥18
* NIHSS ≥ 4
* ICA or M1 or M2 MCA occlusion on pre-thrombectomy MRA or CTA
* Onset (last-seen-well) time to randomization time within 24 hours
* Pre-stroke modified Rankin Scale≤ 3.
* Patient ineligible for IV tPA, per national AHA/ASA Guidelines.
* Having undergone endovascular thrombectomy with less than a complete reperfusion (<TICI 2c, 3) for receiving post-thrombectomy adjunct C-tDCS.
* Undergoing endovascular thrombectomy, per national AHA/ASA Guidelines for patients who are assigned to pre-thrombectomy bridging session at Tiers 5, 6.
* A signed informed consent is obtained from the patient or patient's legally authorized representative

Exclusion criteria

* Acute intracranial hemorrhage
* Evidence of a large Ischemic core volume (ADC < 620 µm2/s or rCBF< 30%) ≥ 100 ml
* Presence of tDCS contraindications - electrically or magnetically activated intracranial metal and non-metal implants.
* Pregnancy
* Severe contrast allergy or absolute contraindication to iodinated contrast preventing endovascular intervention.
* History of seizure disorder or new seizures with presentation of current stroke
* Evidence of any other major life-threatening or serious medical condition that would prevent completion of the study protocol including attendance at the 3-month follow-up visit
* Concomitant experimental therapy
* Preexisting scalp lesion at the site of the stimulation or presence of skull defects (may alter current flow pattern)
* Preexisting coagulopathy, consist of a platelet count of ≤ 100, INR ≥ 3, PTT ≥ 90.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2019-07-28 (Actual); Primary Completion 2022-04-01 (Actual); Study Completion 2022-04-01 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- University of California- Los Angeles (UCLA), Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Groups:
- Active Stimulation Arm: Patient received 1 mA of high-definition cathodal transcranial direct current for 5 minutes before endovascular procedure (EVT). Patient did not complete the pre-planned 20 minutes of stimulation due to the initiation of EVT.
Period: Overall Study
Arm/Group | Active Stimulation Arm | Sham Arm
Started | 1 | 0
Completed | 0 | 0
Not Completed | 1 | 0

BASELINE CHARACTERISTICS:
Population: Study was stopped early.
Groups:
- Active Stimulation Arm: Patient received 1 mA of high-definition cathodal transcranial direct current for 5 minutes before endovascular procedure (EVT). The pre-planned 20-min stimulation was not completed due to EVT initiation.
- Sham Arm: Patients in the sham stimulation arm were planned to have the cap and electrodes in place but without delivery of electrical stimulation.
  No patient was enrolled in sham arm as the study was stopped early due to slow enrollment rate.
- Total: Total of all reporting groups
Arm/Group | Active Stimulation Arm | Sham Arm | Total
Number analyzed (Participants) | 1 | 0 | 1
Age, Continuous [Mean (Full Range); unit: years] | 95 [95 to 95] |  | 95 [95 to 95]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 |  | 1
  Male | 0 |  | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 |  | 0
  Asian | 0 |  | 0
  Native Hawaiian or Other Pacific Islander | 0 |  | 0
  Black or African American | 1 |  | 1
  White | 0 |  | 0
  More than one race | 0 |  | 0
  Unknown or Not Reported | 0 |  | 0

OUTCOME MEASURES:

1. Primary Outcome: Primary Safety Outcome- Number of Participants With Symptomatic Intracranial Hemorrhage (SICH)
Description: Symptomatic intracranial hemorrhage (SICH) is defined as an increase of 4 or more points on the National Institute of Health Stroke Scale (NIHSS) total score within 24 hours of stimulation associated with parenchymal hematoma type 1 (PH1), parenchymal hematoma type 2 (PH2), remote intraparenchymal hemorrhage (RIH), subarachnoid hemorrhage (SAH), or intraventricular hemorrhage (IVH).
  The NIHSS is a 15-item neurologic examination stroke scale used to evaluate the effect of acute stroke on the levels of consciousness, language, neglect, visual-field loss, extraocular movement, motor strength, ataxia, dysarthria, and sensory loss. A trained observer rates the patent's ability to answer questions and perform activities. Ratings for each item are scored with 3 to 5 grades with 0 as normal, and there is an allowance for untestable items. Accordingly, 0 is the lowest and 42 is the highest total score possible. In the NIHSS, the higher the score, the more impaired a stroke patient is.
Time Frame: At 24-hour post-stimulation
Population: The study was stopped early after the enrollment of the first patient.
Measure: Count of Participants; unit: Participants
Groups:
- Sham Arm: Patients in the sham stimulation arm were planned to have the cap and electrodes in place, but without delivery of electrical stimulation.
  No patient was enrolled in the sham arm as the study was stopped early due to slow enrollment rate.
Arm/Group | Active Stimulation Arm | Sham Arm
Number analyzed (Participants) | 1 | 0
Participants | 0 | 0

2. Primary Outcome: Primary Tolerability Outcome-Number of Participants Completing the Protocol-assigned Stimulation
Description: The percentage of the patients completing the protocol-assigned stimulation treatment with no intolerability.
Time Frame: After 5 minutes of stimulation period
Population: The study was stopped early after the enrollment of the first patient.
Measure: Count of Participants; unit: Participants
Arm/Group | Active Stimulation Arm | Sham Arm
Number analyzed (Participants) | 1 | 0
Participants | 1 |

3. Primary Outcome: Primary Feasibility Outcome- Assessing the Speed of Stimulation Implementation From Randomization.
Description: The median times from randomization to bridging C-tDCS initiation and the time form end of endovascular thrombectomy procedure to adjunctive C-tDCS initiation in the last 10 enrolled patients.
Time Frame: Median time from randomization to tDCS initiation
Population: Study was stopped early after enrollment of first patient. No patient was enrolled in sham arm.
Measure: Number; unit: minutes
Arm/Group | Active Stimulation Arm | Sham Arm
Number analyzed (Participants) | 1 | 0
minutes | 12 |

4. Secondary Outcome: Secondary Safety Outcome-Number of Participants With Asymptomatic Intracranial Hemorrhage (AICH)
Description: AICH is defined as intracranial hemorrhage not associated with National Institute of Health Stroke Scale (NIHSS) total score worsening of ≥ 4.
  The NIHSS is a 15-item neurologic examination stroke scale used to evaluate the effect of acute stroke on the levels of consciousness, language, neglect, visual-field loss, extraocular movement, motor strength, ataxia, dysarthria, and sensory loss. A trained observer rates the patent's ability to answer questions and perform activities. Ratings for each item are scored with 3 to 5 grades with 0 as normal, and there is an allowance for untestable items. Accordingly, 0 is the lowest and 42 is the highest total score possible. In the NIHSS, the higher the score, the more impaired a stroke patient is.
Time Frame: At 24-hour post-stimulation
Population: One patient was enrolled in the Active arm and no patient in sham arm.
Measure: Number; unit: participants
Arm/Group | Active Stimulation Arm | Sham Arm
Number analyzed (Participants) | 1 | 0
participants | 0 |

5. Secondary Outcome: Secondary Safety Outcome-Number of Participants With Early Neurologic Deterioration
Description: Worsening of total score ≥ 4 on NIHSS during the 24-hour period after stimulation, with or without intracranial hemorrhage.
  The NIHSS is a 15-item neurologic examination stroke scale used to evaluate the effect of acute stroke on the levels of consciousness, language, neglect, visual-field loss, extraocular movement, motor strength, ataxia, dysarthria, and sensory loss. A trained observer rates the patent's ability to answer questions and perform activities. Ratings for each item are scored with 3 to 5 grades with 0 as normal, and there is an allowance for untestable items. Accordingly, 0 is the lowest and 42 is the highest total score possible. In the NIHSS, the higher the score, the more impaired a stroke patient is.
Time Frame: At 24-hour post-stimulation
Population: One patient was enrolled in the Active arm and no patient in sham arm.
Measure: Count of Participants; unit: Participants
Arm/Group | Active Stimulation Arm | Sham Arm
Number analyzed (Participants) | 1 | 0
Participants | 0 |

6. Secondary Outcome: Secondary Safety Outcome-Number of Participants With Mortality
Description: Rate of mortality
Time Frame: At 90 days post-stimulation
Population: One patient was enrolled in the Active arm and no patient in sham arm.
Measure: Count of Participants; unit: Participants
Arm/Group | Active Stimulation Arm | Sham Arm
Number analyzed (Participants) | 1 | 0
Participants | 1 |

7. Secondary Outcome: Secondary Safety Outcome-Number of Participants With All Serious Adverse Events (Anticipated and Unanticipated)
Description: A serious adverse event (SAE) is any adverse event that is fatal, is life-threatening, is permanently or substantially disabling, requires or prolongs hospitalization, or requires medical or surgical intervention to prevent one of the above outcomes. Anticipated serious adverse events were defined as SAEs that are expected and related to acute ischemic stroke complications such as headache, stroke recurrence, pneumonia, systemic blood clots, Family withdrawal of care, etc. An unanticipated serious adverse event is an SAE that is not deemed an ischemic stroke complication and adjudicated as possibly related to study treatment.
Time Frame: At 90 days post-stimulation
Population: One patient was enrolled in the Active arm and no patient in sham arm.
Measure: Count of Participants; unit: Participants
Arm/Group | Active Stimulation Arm | Sham Arm
Number analyzed (Participants) | 1 | 0
Participants | 1 |

8. Other Pre Specified Outcome: Exploratory Imaging Efficacy Outcome- Assessing Imaging Biomarker of Neuroprotection and Collateral Enhancement
Description: By comparing the baseline MR/CT imaging with the MR/CT imaging at 2-hour (early) and 24-hour (final) post-stimulation, the following were planned to be measured: 1) Final penumbra salvage proportion, 2) Final hypoperfusion lesion reduction, 3) Early relative quantitative cerebral blood volume (qrCBV) enhancement.
Time Frame: Change in the penumbral volume between the timepoints: baseline, 2- hour, and 24-hour post-stimulation
Population: One patient was enrolled in the Active arm and no patient in sham arm. Secondary outcome data were not collected in the one active patient.
Arm/Group | Active Stimulation Arm | Sham Arm
Number analyzed (Participants) | 0 | 0

9. Other Pre Specified Outcome: Exploratory Clinical Efficacy Outcome- Assessing 3 Months Disability
Description: Examining the clinical outcomes of 3-month modified Rankin Scale.
  The modified Rankin Scale is a commonly used scale for measuring the degree of disability or dependence in the daily activities of people who have suffered a stroke or other causes of neurological disability.The scale runs from 0-6, running from perfect health without symptoms to death.
Time Frame: At day-90 post stimulation
Population: as for outcome 8
Arm/Group | Active Stimulation Arm | Sham Arm
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: 90 days after enrollment
Description: Study was stopped early, no sham was enrolled
Groups:
- Sham Arm: Patients in the sham stimulation arm were planned to have the cap and electrodes in place, but without delivery of electrical stimulation.
  No patient was enrolled in sham arm as the study was stopped early due to slow enrollment rate.
Arm/Group | Active Stimulation Arm | Sham Arm
All-Cause Mortality (participants affected / at risk) | 1/1 | 0/0
Serious Adverse Events (participants affected / at risk) | 1/1 | 0/0
Other Adverse Events (participants affected / at risk) | 0/1 | 0/0
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Active Stimulation Arm (N=1) | Sham Arm (N=0)
Anticipated serious adverse events (Nervous system disorders) | 1 (1) | NA — Anticipated serious adverse events were defined as SAEs that are expected and related to acute ischemic stroke complications such as death related to family withdrawal of care (as in our patient), death due to malignant ischemic stroke, etc.
Unanticipated serious adverse event (Nervous system disorders) | 0 (0) | NA — An unanticipated serious adverse event is an SAE that is not deemed an ischemic stroke complication and adjudicated as possibly related to study treatment

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-01-12): https://cdn.clinicaltrials.gov/large-docs/77/NCT04061577/Prot_SAP_000.pdf
  • Informed Consent Form (2021-04-27): https://cdn.clinicaltrials.gov/large-docs/77/NCT04061577/ICF_001.pdf